CLINICAL TRIAL: NCT02988596
Title: Management and Treatment of Sport-related Concussion: Early Multidimensional Rehabilitation Versus Enhanced Graded Exercise
Brief Title: Role of Rehabilitation in Concussion Management: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Medical College of Wisconsin (Other); National Football League Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1228
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Concussion, Brain
Keywords: Concussion; Rehabilitation
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Graded Exertion (Active Comparator): At the time of the injury, participants will be given guided activity instructions regarding what activities to consider and how to observe for increases in symptoms. The focus will be on guided activity and not on restriction. Symptoms will be assessed at the end of each day. Once the patient has been asymptomatic for 24 hours or within 85% of their baseline symptom score (BSS) they will begin the enhanced graded exertion progression (Zurich/Berlin protocol). This protocol will follow the Zurich/Berlin guidelines, but will be enhanced to include sports and skill specific activities. Each step will be completed on a separate day. A medical professional will determine the symptom status of the athlete and when the graded exertion will begin.
  Interventions: Other: Enhanced Graded Exertion
- Multidimensional Active Rehabilitation (Experimental): At injury, participants are given instructions regarding guided activities to consider and how to observe for symptom increase. Focus is on guided activity, not restriction. The intervention consists of 5 phases designed to facilitate an active approach to concussion rehabilitation. Phases are symptom stabilization, impairment reduction, activity integration, recovery acceleration, and sport specific application. Participants complete phase specific activities under direction of a clinical professional, and progress upon meeting specific requirements. Participants are required to spend at least 2 days in Phase 1; subsequent phases are completed on separate days. Once asymptomatic for 24 hours or within 85% of their BSS they begin the enhanced graded exertion progression (Zurich/Berlin protocol).
  Interventions: Other: Multidimensional Active Rehabilitation

INTERVENTIONS:
Other: Multidimensional Active Rehabilitation — Participants will be asked to complete activities aimed at: stabilization of symptoms, impairment reduction, activity integration, recovery acceleration and sport specific application during a 20 minute session at least 4 times a week. Activities will be selected by the supervising clinician with respect to the specific impairment presentation of each participant. Session logs will be completed by each clinician and will include the following information: initial symptom checklist, activity parameters, percentage of rest during the session, participants rating of perceived exertion, and final symptom checklist, session satisfaction rating, and session feedback.
  Arms: Multidimensional Active Rehabilitation
Other: Enhanced Graded Exertion — Participants will be asked to use their symptoms to guide their activity from the time of their injury until they are asymptomatic. Once they are asymptomatic they will begin the graded exertion (Zurich/Berlin Protocol). During this time clinicians will complete session logs that include the following information: initial symptom checklist, phase of graded return to play progression, activity parameters, percentage of rest during the session, participants rating of perceived exertion, and final symptom checklist, session satisfaction rating, and session feedback.
  Arms: Enhanced Graded Exertion

SUMMARY:
Approximately 420 professional and amateur athletes will participate in rehabilitation during recovery after sports-related concussion. Participants will be cluster randomized, by study site, to a specific study arm. Participants will complete post-injury assessments and the intervention of their randomized group aimed at understanding the effects of a multidimensional rehabilitation protocol versus enhanced graded exertion on clinical recovery, return to play, and patient outcomes after sport related concussion

DETAILED DESCRIPTION:
Approximately 6,600 athletes will complete baseline assessments and 420 of these individuals who suffer a concussion during the course of study will be directed through the post-injury protocol. Following injury, participants will complete post-injury assessments and follow the specific intervention of their randomized group. Post-injury assessments will focus on the following: postural stability, neuro-cognitive function, symptom presence and severity, fatigue, vision, dual-task ability, and mental status. Participants will complete outcome assessments at the following time points: time of injury, 24-48 hours post-injury, asymptomatic, and one month post return to play. Symptoms and physical and cognitive activity will be assessed daily from the first assessment point to 7 days post return to play. Session logs will be kept by the supervising clinician at each study site regardless of study arm. Baseline and outcome assessments will be entered into a secure online platform, each study site will have the option for paper records of outcomes and session logs to be double entered into the electronic system at a later date.

ELIGIBILITY:
Subjects will be recruited from 3 cohorts of athletes: 1) high school; 2) college/university and 3) professional.

HIGH SCHOOL COLLEGE/UNIVERSITY COHORTS:

Inclusion criteria:

* Individuals who are at least 13 years of age and a rostered student-athlete on the participating teams at the enrolled schools (football, wrestling, men's/women's soccer, men's/women's lacrosse, and men's/women's ice hockey, men's/women's rugby, and men's/women's basketball or other sports designated at the site).

Exclusion criteria:

* Individuals who are at least 13 years of age and those not rostered in a sport at his/her school.

PROFESSIONAL COHORT:

Inclusion criteria:

* Individuals who are 18 years of age or older and rostered on one of the participating professional teams.

Exclusion criteria:

* Individuals under 18 years of age and those not rostered on one of the participating professional teams.

ELIGIBILITY FOR THE STUDY INTERVENTION: ALL COHORTS

Inclusion criteria:

* Only those athletes with a concussion, guided by the following definition will engage in their respective intervention arms following concussion. The study definition is one from the Department of Defense (DOD). This definition was chosen, as it is s a guiding definition in the NCAA-DOD grand alliance Concussion Assessment, Research and Education (CARE) consortium, the largest concussion study to date (http://www.careconsortium.net/about/).
* Concussion will be defined as a change in brain function following a force to the head, which may (or may not) be accompanied by temporary loss of consciousness (LOC) (if LOC, temporary is study defined as < 30 minutes based on the Mayo traumatic brain injury (TBI) severity guidelines), but is identified in awake individuals with measures of neurologic and cognitive dysfunction, as indicated by 1 or more the symptoms listed below.

Symptoms: headache, 'pressure in the head', neck pain, nausea/vomiting, dizziness, blurred vision, balance problems, sensitivity to light, sensitivity to noise, feeling slowed down, felling like 'in a fog', 'don't feel right, difficulty concentrating, difficulty remembering, fatigue/low energy, confusion, drowsiness, trouble falling asleep, more emotional, irritability, sadness, nervous/anxious.

* These symptoms are from the international consensus document on concussion in sport and represent the most common 22 symptoms of concussion (McCroy & Concussion in Sport Group, 2013). All concussions are, by general definition, mild TBIs with Glasgow Coma Score (GCS) scores of 13-15 (with the majority being 14-15). No athlete with a GCS <13 will be started in the intervention progression of either arm.

Exclusion criteria:

* Individuals with any positive/abnormal clinical neuroimaging finding(s) following injury WILL NOT enter the intervention or will discontinue the intervention should these findings be observed after intervention has begun.
* In addition, any individual presenting with any of the moderate-severe TBI presentation as defined in the Mayo definitions (Malec, 2007) will not enter the intervention or will be withdrawn if observed at a later time. Although these individuals will be discontinued from the intervention, the investigators will continue to collect assessment time point data on these individuals and documentation for their overall care.

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Average Days to Recovery | 1 to approximately 240 days
  Average number of days from injury to recovery (recovery is defined as full clearance by physician for full return to sport participation)

SECONDARY OUTCOMES:
Change in Fatigue from Baseline to 1 Month Post Return to Play | Baseline, 24-48 hrs post injury, asymptomatic (1 to approximately 240 days), 1 month post return to play
  Participants are asked to rate their level of fatigue on a scale from 0 (completely exhausted) to 100 (completely alert).
Change in Quality of Life Perception (PROMIS) from Baseline to 1 Month Post Return to Play | Baseline, asymptomatic (1 to approximately 240 days), 1 month post return to play
  The investigators will utilize the short version of the PROMIS general scale and the PROMIS cognitive and fatigue modules. For the PROMIS general scale and modules, participants are asked to rate items on scale from 1-5, each item rating in a given scale is summed and a scale score is computed using PROMIS guidelines.
Change in Concussive Symptoms using the Sport Concussion Assessment Tool (SCAT 3) from Baseline to 1 Month Post Return to Play | Baseline, time of injury (within 6 hrs), 24-48 hrs post injury, asymptomatic (1 to approximately 240 days), 1 month post return to play
  The SCAT 3 concussion symptom checklist is a commonly used symptom assessment following concussion. Participants are asked to rate the severity of 22 symptoms on a scale from 0 (none) to 6 (severe). Each symptom item is added together to compute overall symptom burden.
Change in Psychological Distress using the Brief Symptom Inventory-18 (BSI-18) from Baseline to 1 Month Post Return to Play | Baseline, 24-48 hrs post injury, asymptomatic (1 to approximately 240 days), 1 month post return to play
  The BSI-18 asks the participant to rate their level of distress associated with 18 symptom items on a scale from 0 (not at all) to 4 (extremely), ratings from each item are added together to compute overall symptom distress.
Change in Cognitive Status using the Standard Assessment of Concussion (SAC) from Baseline to 1 Month Post Return to Play | Baseline, time of injury (within 6 hrs), 24-48 hrs post injury, asymptomatic (1 to approximately 240 days), 1 month post return to play
  The SAC will be used to assess cognitive status after acute injury. The SAC has demonstrated validity, reliability, and sensitivity to concussion. The SAC contains sections on orientation, immediate memory, concentration, and delayed memory sections. The sum scores for each of these sections are used to calculate a SAC total score.
Change in Balance using the Balance Error Scoring System (BESS) from Baseline to 1 Month Post Return to Play | Baseline, time of injury (within 6 hrs), 24-48 hrs post injury, asymptomatic (1 to approximately 240 days), 1 month post return to play
  The Balance Error Scoring System (BESS) is a commonly used measure of static balance and postural stability. A combination of three stances (narrow double leg stance, single leg stance, and tandem stance) and two footing surfaces (firm surface/floor or medium density foam) are used for the test. Each stance is held, with hands on hips and eyes closed, for 20 seconds. Points are given for specific behaviors ("errors"), including opening eyes, lifting hands off hips, or stepping, stumbling, or falling. It will be conducted by a trained study team member. Safety issue: Fall related injuries.
Change in Cognition from Baseline to 1 Month Post Return to play | Baseline, 24-48 hrs post injury, asymptomatic (1 to approximately 240 days), 1 month post return to play
  Computerized neuropsychological testing to determine cognitive functioning will be utilized. Percentiles of participant's overall achievement on the computerized neurocognitive test is reported. Measures will include Immediate Postconcussion and Cognitive Test (ImPact) and Concussion Vital Signs (CVS) and CogState (Axon Sports).
Change in Near-Point Convergence from Baseline to 1 Month Post Return to Play | Baseline, 24-48 hrs post injury, asymptomatic (1 to approximately 240 days), 1 month post return to play
  Near-point convergence is a commonly used oculomotor exam that defines the amplitude of convergence or the closest point in space where the patient can hold fusion, and therefore, see one target. Participants complete 3 trials assessing near-point convergence: the average of the three trials is recorded.
Change in Dual-Task Ability using a Gait + Digit Span Dual-Task from Baseline to 1 Month Post Return to Play | 24-48 hrs post injury, asymptomatic, (1 to approximately 240 days) 1 month post return to play
  The Gait + Digit Span Dual-Task begins with a walking task of 7 meters (timed). The participant then completes a memory recall task and is assessed for accuracy. Finally, the participant is asked to complete these two tasks simultaneously while the clinician records the same measures. Safety issue: Fall related injury. All Dual-Task testing will be supervised by a clinical professional or physician.
Change in Daily Concussion Symptoms | Daily post injury - 1 to approximately 240 days
  Participants are asked to complete a modified version of the SCAT 3 to assess symptom burden.
Change in Daily Activity | Daily post injury - 1 to approximately 240 days
  Participants are asked to complete a cognitive and physical daily activity log to assess cognitive and physical activity burden.

CONTACTS AND LOCATIONS:
Overall Officials: Johna K Mihalik, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (11):
- United States (7):
  - North Carolina Central University, Durham, North Carolina
  - Elon University, Elon, North Carolina
  - Orange County High School, Hillsborough, North Carolina
  - Northwood High School, Pittsboro, North Carolina
  - Catawba College, Salisbury, North Carolina
  - Lynchburg College, Lynchburg, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - York University, Toronto, Ontario
  - Canadian Football League, Toronto, Ontario
- New Zealand Rugby, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malec JF, Brown AW, Leibson CL, Flaada JT, Mandrekar JN, Diehl NN, Perkins PK. The mayo classification system for traumatic brain injury severity. J Neurotrauma. 2007 Sep;24(9):1417-24. doi: 10.1089/neu.2006.0245. PMID 17892404
- [Derived] Register-Mihalik JK, Guskiewicz KM, Marshall SW, McCulloch KL, Mihalik JP, Mrazik M, Murphy I, Naidu D, Ranapurwala SI, Schneider KJ, Gildner P, Salmon DM, Auton B, Bowman TG, Hall EE, Hynes LM, Jewell E, Ketcham CJ, Siler CW, Sullivan SJ, Kostogiannes V, McCrea MA; Active Rehab Study Consortium. Symptom Exacerbation and Adverse Events During a Randomized Trial of Early-Stage Rehabilitation After Sport-Related Concussion: Safety Outcomes From the Active Rehab Study. J Athl Train. 2024 Dec 1;59(12):1163-1170. doi: 10.4085/1062-6050-0696.23. PMID 38775119
- [Derived] Register-Mihalik JK, Guskiewicz KM, Marshall SW, McCulloch KL, Mihalik JP, Mrazik M, Murphy I, Naidu D, Ranapurwala SI, Schneider K, Gildner P, McCrea M; Active Rehab Study Consortium Investigators. Methodology and Implementation of a Randomized Controlled Trial (RCT) for Early Post-concussion Rehabilitation: The Active Rehab Study. Front Neurol. 2019 Nov 8;10:1176. doi: 10.3389/fneur.2019.01176. eCollection 2019. PMID 31781021